CLINICAL TRIAL: NCT06299436
Title: Hemodynamic Assessment of underLying myocyTe Function in Right Heart Failure
Acronym: HALT-RHF
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00426760; R01HL172830 (NIH)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Pulmonary Hypertension; Right Heart Failure Due to Left Heart Failure
Keywords: right heart failure; heart failure; cardiomyopathy; pulmonary hypertension; heart failure with reduced ejection fraction
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (plasma and serum); right ventricular endomyocardial biopsy specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Right ventricular (RV) failure is recognized to worsen patient outcomes in the setting of heart failure with reduced ejection fraction (HFrEF)-related pulmonary hypertension (PH), yet the investigators fall short in trying to identify and treat it. The current proposal will (1) determine the best clinical indicators of intrinsic RV myocyte contractile failure in humans with HFrEF-PH, (2) clarify underlying mechanisms, and (3) test novel treatments on RV myocytes. The long-term goal of this proposal will be to better identify and treat RV failure in humans suffering from HFrEF-PH.

DETAILED DESCRIPTION:
This proposal aims to improve diagnosis and mechanistic understanding of right ventricular (RV) myocyte dysfunction in heart failure patients with reduced ejection fraction and pulmonary hypertension (HFrEF-PH). RV dysfunction is common and hastens poor outcomes in HFrEF-PH. Despite its importance, clinical ability to characterize it remains imprecise. This frustrates prognostic and therapeutic efforts in many scenarios, such as the prediction of RV failure following left ventricular assist device. In 2023, the investigators reported that RV myocyte contractile reserve indices, such as calcium-activated isometric tension and length-dependent active tension, are reduced in RV tissue of explanted end-stage human HFrEF-PH hearts. Notably, clinical indices correlated modestly with calcium-activated tension but completely failed to capture depression of length-dependent tension, the latter a key contributor to RV Frank-Starling reserve. This deficiency highlights one possible reason why clinical indices fail to identify RV failure. A shortcoming of this work was its study of end-stage disease, and the investigators believe better clinical correlates of myocyte dysfunction from earlier-stage disease may provide more insight at a time point when interventions would still be helpful. The investigators central hypothesis is that clinical identification of RV myocyte disease in HFrEF-PH requires measuring RV contractile reserve, as is elicited during exercise. The investigators prior study of primary PH patients supports this, and new preliminary data in patients with PH secondary to heart failure does so as well. Delving deeper, the investigators recently reported a novel deficiency of the sarcomere thick filament in HFrEF-PH RV myocytes, driven by an excess of myosin in the inactive super-relaxed state that hinders its recruitment to form cross-bridges by either calcium- or stretch-activation. The latter is important as it is not seen in small rodents, and only recently reported in pigs, thus newly linking super-relaxed myosin to RV myocyte and chamber reserve in humans. The investigators new phospho-proteomic data shows less myosin binding protein-C phosphorylation yet more phosphorylation of several sarcomere Z-disc proteins, and supports the potential role based on kinase and phosphatase modifications.

This proposal was spawned by these recent findings. The investigators objectives are to: (1) identify clinical indices that capture RV myocyte reserve failure in earlier-to-mid stage HFrEF-PH; (2) uncover mechanisms of myocyte length-dependent contractile depression; and (3) test sarcomere-activating drugs that might prove useful for HFrEF-PH RV failure. The investigators combine state-of-the-art pressure-volume loop and clinical assessments of RV chamber function with phenotyping of the myocyte contractile apparatus. The investigators further explore a new role of super-relaxed myosin in depressed myocyte reserve. The proposal leverages my translational and basic muscle expertise developed over the past several years with K23 support, and a stellar collaborative team. Its objectives align with NHLBI strategic visions for the RV and advanced HF. There are three Specific Aims:

Aim 1. Test whether clinical measures of RV exercise reserve better reflect RV myocyte contractile dysfunction in earlier-stage HFrEF-PH. HFrEF patients referred for right heart cath undergo a well-established protocol at Johns Hopkins to assess clinical hemodynamic and echocardiographic RV indices alongside RV pressure-volume loop parameters at rest and with supine bicycle exercise. RV endomyocardial biopsies are obtained, and isolated myocytes permeabilized to assess contractile mechanics and calcium- and length-activated tension. The investigators then test whether clinical RV exercise reserve parameters will more sensitively reflect RV myocyte contractile reserve limitations than commonly used resting measures of RV function.

Aim 2. Determine roles and identities of phosphorylation mediators of reduced HFrEF-PH RV myocyte length-dependent reserve. New phospho-proteomic data finds protein kinase A (PKA)-hypophosphorylation of thick filament proteins and hyperphosphorylation of Z-disc scaffold proteins in HFrEF-PH RV myocardium. PKA incubation increases myocyte length-dependent tension, while protein phosphatase 2a (which does not reverse PKA changes) improves calcium-activated tension. The investigators test the relevance to myocyte contractile reserve failure in HFrEF-PH in permeabilized RV myocytes by selective kinase and phosphatase incubation, then selectively mutate high-value phospho-modified sites to test the role in length-dependent activation.

Aim 3: Determine whether newer sarcomere-activating drugs restore HFrEF RV myocyte length-dependent tension. Two sarcomere-activating drugs are tested in HFrEF-PH RV myocytes: danicamtiv and CK-136, which should augment length-dependent tension better than similar, previously tested drugs. The investigators determine impact on skinned myocyte contractile reserve, then test if the clinical RV reserve indices identified in Aim 1 can predict impact on individual HFrEF-PH RV myocytes from the same patient.

Expected outcomes: the investigators will identify optimal clinical indices of RV reserve failure in HFrEF-PH, clarify myocyte mechanisms of length-dependent reserve, and test novel RV drugs. Findings will impact RV failure due to HFrEF-PH and should apply to its other causes as well. The investigators research team has exceptional expertise in translational RV phenotyping and muscle biophysics and is uniquely poised to deliver on this proposal.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 90 years of age
* Diagnosed with heart failure with reduced ejection fraction (LV ejection fraction ≤ 40-50%)
* Can safely hold direct oral anticoagulant (DOAC) vitamin K antagonist (VKA) for 48 hours prior to the procedure

Exclusion Criteria:

* Unable to interrupt VKA anticoagulation
* Point of care International Normalized Ratio (INR) > 1.5
* Pregnant patients
* Acute hospitalization or decompensation within 2 weeks prior to study date
* Participation in a study involving an investigational drug within 4 weeks prior to study date
* Inability to lie flat in the supine position
* Symptomatic hemodynamic instability at rest or during the procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who have heart failure with reduced ejection fraction, defined by a left ventricular ejection fraction less than or equal to 40-50%.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy based on Area Under Curve (AUC) | 5 years
  Diagnostic accuracy (AUC), as determined by combination of sensitivity and specificity, of multiple clinical metrics will be compared to determine which best identifies underlying right ventricular myocyte contractile dysfunction.

SECONDARY OUTCOMES:
Percentage improvement in ex vivo right ventricular tissue sample | 5 years
  Percentage improvement is defined as the percent difference in ex vivo right ventricular tissue sample myocyte contractility before and after experimental exposure to sarcomere-activating agent. Note this testing occurs on tissue samples, not in human subjects.
Predictive capacity (based on likelihood ratio) | 5 years
  Combining primary and secondary outcomes, the predictive capacity of clinical metrics will be determined for anticipating a response to sarcomere-activating agent.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hsu, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No